CLINICAL TRIAL: NCT05107999
Title: Stigma and Efficacy of Zhizhu Kuanzhong Capsules Versus Doxepin in the Treatment of Refractory Functional Dyspepsia: a Randomized Controlled Trial
Brief Title: Stigma and Efficacy of Zhizhu Kuanzhong Capsules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, professor, chief physician, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJYYTCM
Record Dates: First submitted 2021-09-26; First posted 2021-11-04 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Functional Gastrointestinal Disorders; Dyspepsia; Psychosomatic Disorder
MeSH Terms: conditions — Gastrointestinal Diseases; Dyspepsia; Psychophysiologic Disorders | interventions — Medicine, Chinese Traditional; Doxepin; Neurotransmitter Agents; Antidepressive Agents

STUDY DESIGN:
Intervention Model Description: Zhizhu Kuanzhong (ZZKZ) group was treated with ZZKZ capsules with omeprazole. Antidepressant group was treated with doxepin with omeprazole.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zhizhu Kuanzhong（ZZKZ） group (Experimental): Patients in ZZKZ group were given ZZKZ (2 capsules tid) plus omeprazole (20 mg bid). ZZKZ was applied after each meal. Omeprazole was applied twice daily, before breakfast and supper.
  Interventions: Drug: Zhizhu Kuanzhong capsules (ZZKZ)
- Doxepin group (Active Comparator): Patients in doxepin group were given doxepin (25 mg tid) plus omeprazole (20 mg bid). Doxepin was applied after each meal. Omeprazole was applied twice daily, before breakfast and supper.
  Interventions: Drug: Doxepin Hydrochloride (Doxepin)

INTERVENTIONS:
Drug: Zhizhu Kuanzhong capsules (ZZKZ) — FD patients were treated with ZZKZ and omeprazole for 4 weeks.
  Other Names: Traditional Chinese medicine
  Arms: Zhizhu Kuanzhong（ZZKZ） group
Drug: Doxepin Hydrochloride (Doxepin) — FD patients were treated with doxepin and omeprazole for 4 weeks.
  Other Names: Neuromodulators; Antidepressants
  Arms: Doxepin group

SUMMARY:
Antidepressants are effective in patients with functional dyspepsia (FD), however, the stigma related with FD and antidepressants could affect treatment adherence and efficacy. Zhi Zhu Kuan Zhong capsules (ZZKZ), a traditional Chinese medicine fomula, showed therapeutic potential for FD. The study was designed to investigate whether ZZKZ could alleviate stigma in FD and obtain identical effects in patients with refractory FD.

DETAILED DESCRIPTION:
Patients with dyspepsia have poor quality of life and emotional distress. The pathophysiology of FD is complex and multifactorial, including factors related to central nervous system and peripheral sensory system. Abundant drugs have been trialed to treat FD patients, but the treatment options remain limited and far from optimal. Antidepressants were beneficial in the treatment of FD. But the antidepressant prescriptions often aggravate the stigma of patients with FD, hinder doctor-patient communication, and reduce treatment compliance. Some patients with strong stigmatized feelings towards antidepressants refused to take the medications, and stigma related with antidepressants could ultimately affect the efficacy of FD. Zhizhu Kuanzhong capsules (ZZKZ), a commonly used traditional Chinese medicine (TCM) formula, had shown effectiveness in relieving dyspeptic symptoms. It has a long culture and history in promoting the function of brain and GI tract in whole, which is widely accepted by populations who were familiar with TCM. The study was designed to observe whether ZZKZ could alleviate stigma of patients and obtain identical effects in patients with FD, therefore provide a new insight in the treatment of FD.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria includes:
* 18-70 years old;
* education level higher than middle school;
* met the Rome IV criteria for FD;
* absence of abnormalities on physical examination, laboratory tests (including a routine blood test, blood glucose, and liver function examination), and abdominal imaging and GI endoscopy within 6 months;
* absence of Helicobacter pylori infection;
* signed written informed consent for participation in the study.

Exclusion Criteria:

* The exclusion criteria includes:
* evidence of organic digestive diseases;
* diabetes, cancer and other diseases might affect GI function;
* pregnancy, lactation or breastfeeding;
* a history of allergic reaction to any of the drugs used in the study;
* participation in other clinical trials in the previous 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Leeds Dyspepsia Questionnaire (LDQ) scores at 4 weeks from baseline were obtained to assess the dyspepsia condition after treatment. | 4 weeks
  The LDQ scores of 0-4 were classified as very mild dyspepsia, 5-8 as mild dyspepsia, 9-15 as moderate dyspepsia, and >15 as severe or very severe dyspepsia.
Changes of Patient Health Questionnaire-9 (PHQ-9) scores at 4 weeks from baseline were obtained to assess the depression condition after treatment. | 4 weeks
  The PHQ-9 scores of 0-4 were classified as none or minimal depression, 5-9 as mild, 10-14 as moderate, 15-19 as moderately severe, and ≥20 as severe depression.
Changes of Generalized Anxiety Questionnaire-7 (GAD-7) scores at 4 weeks from baseline were obtained to assess the anxiety condition after treatment. | 4 weeks
  The GAD-7 scores of 0-4 were classified as the absence of anxiety, 5-9 as mild, 10-14 as moderate, and ≥15 as severe.

SECONDARY OUTCOMES:
Changes of Internalized stigma scale (ISS) scores at 4 weeks from baseline were obtained to assess the internalized stigma of patients after treatment. | 4 weeks
  The Internalized stigma scale (ISS) is a 24-item self-report questionnaire with items ranked on a 4-point Likert scale (strongly disagree = 1 to strongly agree = 4 points). The ISS scores are calculated by summing the values for each item and dividing by the number of questions answered for each scale. Higher scores indicate higher levels of ISS. The ISS scores of 1-2 were classifies as minimal, 2-2.5 as mild, 2.5-3 as moderate, 3-4 as severe.
Changes of Perceived stigma scale (PSS) scores at 4 weeks from baseline were obtained to assess the perceived stigma of patients after treatment. | 4 weeks
  The Perceived stigma scale (PSS) is a 10-item questionnaire with items ranked on a 5-point Likert scale (seldom = 1 to always = 5 points). The scores are calculated by summing the values for each item and dividing by the number of questions answered for each scale. Minimum to maximum score is 1 to 5 points. Higher scores indicate higher levels of PSS. The PSS scores of 1-2 were classifies as minimal, 2-3 as mild, 3-4 as moderate, 4-5 as severe.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Liang Chen, PhD, Principal Investigator — Division of Gastroenterology and Hepatology, Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xiao Y, Li Y, Shu J, Li Y, Xu J, Ren J, Liu D, Wang J, Zhou L, Li Y, Tang G, Tian D, Zhang S, Hou X, Wang H, Li Z, Lv N, Chen M. The efficacy of oral Zhizhu Kuanzhong, a traditional Chinese medicine, in patients with postprandial distress syndrome. J Gastroenterol Hepatol. 2019 Mar;34(3):526-531. doi: 10.1111/jgh.14467. Epub 2018 Oct 12. PMID 30207000
- [Result] Gwee KA, Holtmann G, Tack J, Suzuki H, Liu J, Xiao Y, Chen MH, Hou X, Wu DC, Toh C, Lu F, Tang XD. Herbal medicines in functional dyspepsia-Untapped opportunities not without risks. Neurogastroenterol Motil. 2021 Feb;33(2):e14044. doi: 10.1111/nmo.14044. Epub 2020 Nov 30. PMID 33258198
- [Result] Yan XJ, Luo QQ, Qiu HY, Ji CF, Chen SL. The impact of stigma on medication adherence in patients with functional dyspepsia. Neurogastroenterol Motil. 2021 Feb;33(2):e13956. doi: 10.1111/nmo.13956. Epub 2020 Jul 27. PMID 33184967
- [Result] Feingold JH, Drossman DA. Deconstructing stigma as a barrier to treating DGBI: Lessons for clinicians. Neurogastroenterol Motil. 2021 Feb;33(2):e14080. doi: 10.1111/nmo.14080. Epub 2021 Jan 23. PMID 33484225
- [Result] Holtmann G, Talley NJ. Herbal medicines for the treatment of functional and inflammatory bowel disorders. Clin Gastroenterol Hepatol. 2015 Mar;13(3):422-32. doi: 10.1016/j.cgh.2014.03.014. Epub 2014 Mar 25. PMID 24674944
- [Result] Black CJ, Drossman DA, Talley NJ, Ruddy J, Ford AC. Functional gastrointestinal disorders: advances in understanding and management. Lancet. 2020 Nov 21;396(10263):1664-1674. doi: 10.1016/S0140-6736(20)32115-2. Epub 2020 Oct 10. PMID 33049221